CLINICAL TRIAL: NCT01202968
Title: Effect of Pre-emptive Transcutaneous Neuro-muscular Electrical Stimulation for Dysphagia in Long Term Intubated Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Clinical Associate Professor, Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: chhwang2
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Deglutition Disorder
Keywords: intubation electric stimulation deglutition disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Transcutaneous neuro-muscular electrical stimulation — Neuro-muscular electrical stimulation with two pairs of surface electrodes was applied to submental area. One paired electrodes to be placed horizontally was attached on the anterior half of area between mandible and hyoid bone. The other was affixed to posterior half of the same area far laterally. Bipolar electrical stimulation with pulse rate of 80-Hz, duration of 700 µs and intensity to evoke visible muscle contraction was performed for 60 minutes a day until one day before extubation.
  Other Names: VitalStim (DJO Incorporated, California, USA)

SUMMARY:
It was well known that long term intubation caused a various kind of abnormal presentations of dysphagia such as the increased aspiration risk, the decreased gag reflex, mucosal pathology, the airway stenosis and so on. It was thought that the freezing and impaired proprioception to be developed as a result of dis-use around the pharynx and the larynx while intubation was one of the reason.

Preemptive swallowing manual stimulation applied on the oral cavity to avoid the vicious cycle of dis-use was reported to improve dysphagia after extubation.

Neuromuscular electrical stimulation have been utilized for a wide variety of dysphagia of multiple causes of neuro-muscular disorder.

Supposing that preemptive transcutaneous neuromuscular electrical stimulation to be delivered to the muscles of being involved in swallowing could decrease the degree of dis-use during intubation so that it could reduce the occurence and severity of dysphagia developed after extubation, the investigators plan to perform randomized prospective double blind placebo controlled clinical interventional study.

ELIGIBILITY:
Inclusion Criteria:

* patients to be admitted to the ICU due to the respiratory failure and intubated for at least 48 hours

Exclusion Criteria:

* Past history of intubation
* Past history or current status of traumatic brain injury
* Past history or current status of symptomatic stroke
* Past history or current status of injury of cranial nerves
* Past history or current status of neuromuscular disorder
* Patient not to be expected to be extubated
* Patient to reject the participation
* current usage of neuro-muscular blockers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
oro-pharyngeal swallowing efficiency | as soon as patient could tolerate videofluoroscopic swallowing study after extubation; average of 5 days
  oro-pharyngeal swallowing efficiency was calculated by using the data derived from videofluoroscopic swallowing study

SECONDARY OUTCOMES:
oral transit time | as soon as patient could tolerate videofluoroscopic swallowing study after extubation; average of 5 days
  oral transit time was measured through videofluoroscopic swallowing study
pharyngeal transit time | as soon as patient could tolerate videofluoroscopic swallowing study after extubation; average of 5 days
  pharyngeal transit time was measured through videofluoroscopic swallowing study
oro-pharyngeal transit time | as soon as patient could tolerate videofluoroscopic swallowing study after extubation; average of 5 days
  oro-pharyneal transit time was calculated by using the data derived from videofluoroscopic swallowing study
swallowed volume | as soon as patient could tolerate videofluoroscopic swallowing study after extubation; average of 5 days
  swallowd volume was measured through videofluoroscopic swallowing study
aspiration volume | as soon as patient could tolerate videofluoroscopic swallowing study after extubation; average of 5 days
  aspiration volume was measured through videofluoroscopic swallowing study
presence of aspiration | as soon as patient could tolerate videofluoroscopic swallowing study after extubation; average of 5 days
  presence of aspiration was checked through videofluoroscopic swallowing study
presence of silent aspiration | as soon as patient could tolerate videofluoroscopic swallowing study after extubation; average of 5 days
  presence of silent aspiration was checked through videofluoroscopic swallowing study
penetration-aspiration scale | as soon as patient could tolerate videofluoroscopic swallowing study after extubation; average of 5 days
  penetration-aspiration scale was scored through videofluoroscopic swallowing study

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Study Director — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea